CLINICAL TRIAL: NCT06768996
Title: The Impact of a Caregiver-patient Music Intervention on Social Attention and Connectedness in Persons Living With bvFTD and AD
Brief Title: Music, Social Attention, and Dementia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-40419; T32AG078115 (NIH)
Record Dates: First submitted 2024-12-05; First posted 2025-01-10 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Frontotemporal Dementia; Alzheimer Disease
MeSH Terms: conditions — Frontotemporal Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Control-treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solo Rhythm Production (Active Comparator): Participants randomized to the control condition will complete the same rhythm conditions to the same recorded audio tracks described in the experimental condition. However, they will not interchange their tapping with their caregiver. They will participate in the rhythm task as a solo producer.
  Interventions: Behavioral: Solo Rhythm Production
- Synchronous Rhythm Production (Experimental): The treatment group will take part in a dyad-based musical rhythm production activity facilitated by a trained musician. This activity will involve two rhythm conditions. The first condition requires tapping along to one pre-recorded audio track composed of an ensemble of Brazilian percussion instruments. The second condition requires tapping along with prerecorded audio tracks of rhythms progressively increasing in difficulty. Participants who indicate proficiency in learning to tap along in both conditions will be able to progress to more complex rhythms. All tapping data will be gathered through a Roland digital hand percussion controller.
  Interventions: Behavioral: Synchronous Rhythm Production

INTERVENTIONS:
Behavioral: Synchronous Rhythm Production — The treatment group will take part in a dyad-based musical rhythm production activity facilitated by a trained musician. This activity will involve two rhythm conditions. The first condition requires tapping along to one pre-recorded audio track composed of an ensemble of Brazilian percussion instruments. The second condition requires tapping along with prerecorded audio tracks of rhythms progressively increasing in difficulty. Participants who indicate proficiency in learning to tap along in both conditions will be able to progress to more complex rhythms. All tapping data will be gathered through a Roland digital hand percussion controller.
  Arms: Synchronous Rhythm Production
Behavioral: Solo Rhythm Production — Participants randomized to the control condition will complete the same rhythm conditions to the same recorded audio tracks described in the experimental condition. However, they will not interchange their tapping with their caregiver. They will participate in the rhythm task as a solo producer.
  Arms: Solo Rhythm Production

SUMMARY:
This is an exploratory mixed-methods control-treatment study to evaluate if participation in rhythmic musical activities improves social attention and connectedness in individuals living with mild to moderate bvFTD and AD, and their caregivers. Secondary objectives include evaluating the potential relationships between brain networks associated with rhythm production, social attention, and connectedness in these populations.

DETAILED DESCRIPTION:
The proposed research will evaluate potential relationships between synchronous rhythm production, social attention, and connectedness in persons living with mild to moderate bvFTD and AD and their caregivers. To evaluate these relationships, the proposed research will include data collection and analysis of the following: 1) pre-post evaluation of social attention and connectedness in individuals living with dementia and their caregivers; 2) control-treatment participation in a synchronous (treatment) or solo (control) rhythm production activity; and 3) secondary analysis of structural and functional MRI of resting state network connectivity between networks of the brain including areas associated with rhythm perception and production, namely the fronto-parietal, executive control, sensorimotor, dorsal and ventral attention networks.

ELIGIBILITY:
Inclusion (patients)

* Male or female ≥ 55 years of age living with bvFTD; or ≥ 70 years of age living with AD.
* Documentation of a bvFTD or AD diagnosis as evidenced by one or more known clinical features.
* Written informed consent obtained from subject.

Inclusion (caregivers)

* Male or female ≥ 55 years of age living without diagnosis of neurological or psychiatric disease.
* Individual capable of independent execution of activities of daily living, including personal care and hygiene, dressing, eating, use of a toilet, and mobility.
* Written informed consent.

Exclusion (patients)

* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* community-dwelling individuals not living with bvFTD

  * community-dwelling individuals with normal cognitive functioning
  * Individuals living with Alzheimer's disease or related dementias (primary progressive aphasia, semantic variant FTD, Lewy body dementia, vascular dementia, Parkinson's disease, or mixed dementia)
* Individuals with a score of 2 or higher on the CDR
* Individuals with a history of neuropsychiatric illness that would interfere with performance (e.g., transient psych hx of depression okay, hx of schizophrenia will be excluded) or medicated depression to control symptoms.
* Individuals with unstable (e.g., cancer other than basal cell skin) or chronic (e.g., severe diabetes) medical conditions
* Individuals with MRI contraindications (e.g., pregnancy, claustrophobia, metal implants that are contraindicated for MRI)
* Individuals with physical impairment(s) precluding motor response
* Individuals with inability to walk two blocks without stopping
* Individuals with hearing or vision deficits that will not allow for completion of testing; inability to hear conversation conducted at an average volume (~60 dB)
* Individuals who practice music making or production for at least 30-mins per week

  * This may include instrumental or vocal, writing or arranging, alone or in groups
  * Listening to music for more than 30-mins weekly will not exclude the individual from the study

Exclusion (Caregivers)

* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Community-dwelling individuals living with diagnosis of a neurological or psychiatric disease

  o Community-dwelling individuals with abnormal cognitive functioning
* Individuals living with dementia
* Individuals with a history of neuropsychiatric illness that would interfere with performance (e.g., transient psych hx of depression okay, hx of schizophrenia will be excluded) or medicated depression to control symptoms
* Individuals with unstable (e.g., cancer other than basal cell carcinoma) or chronic (e.g., severe diabetes) medical conditions
* Individuals with physical impairment(s) precluding motor control
* Individuals with inability to walk two blocks without stopping
* Individuals with hearing or vision deficits that will not allow for completion of testing; inability to hear conversation conducted at an average volume (~60 dB)
* Individuals who practice music making or production for at least 30-mins per week

  * This may include instrumental or vocal, writing or arranging, alone or in groups
  * Listening to music for more than 30-mins weekly will not exclude the individual from the study

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Social Attention (TASIT) | Baseline, 2-weeks
  Dependent Variable. Change in social attention will be measured by the TASIT, a 16-item instrument that measures social attention from the care recipient perspective. Items are sectioned by emotion recognition, social inference minimum (sarcasm) or enriched (lies) and assessed using standardized yes-no questions at the end of each section based on four types: think, feel, say, or do.
Degree of rhythmic synchronization between dyad-pairs as determined by autocorrelated inter-tap intervals | Through study completion, an average of one year
  Independent variable. Degree of rhythmic synchronization will be measured via a musical instrument, digital interface (MIDI) and assessed using an automated data analysis tool created explicitly for the purposes of this study.
Caregiver perceived connectedness questionnaire | Baseline, 2-weeks
  A 1-item, 1-7 Likert based scale (1 = very disconnected ... 7 = very connected)
Mutuality Scale | Baseline, 2-weeks
  A 15-item instrument using a 0-4 Likert (0 = not at all … 4 = a great deal) that measures mutuality from the caregiver perspective. Examples include "How close do you feel to the person you care for?" or "How much do you confide in the person you care for?"
Zarit burden | Baseline, 2-weeks
  A 12-item instrument using a 0-4 Likert (0 = never … 4 = nearly always) that measures burden from the caregiver perspective. An example is "Do you feel that your social life has suffered because you are caring for your relative?"
Positive and Negative Experience | Baseline, 2-weeks
  A 12-item instrument using a 1-5 Likert (1 = very rarely or never … 5 = very often or always) that measures an overall affect score that can also be divided into positive and negative feelings. It measures how the participant has felt over the past 4-weeks.
Positive Aspects of Caregiving | Baseline, 2-weeks
  A 9-item instrument using a 1-5 Likert (1 = disagree a lot … 5 = agree a lot) that measures a caregiver's perceptions of their positive experiences in caregiving for their care recipient. An example is "Providing help to [enter name of care recipient] has made me feel more useful."
Trait Empathy (Interpersonal Reactivity Index) | Baseline
  A 28-item instrument using an A-E Likert (A = does not describe me well … E = describes me very well) that measures participants' trait empathic disposition. Four dimensions of trait empathy are used: fantasy scale, empathic concert, perspective taking, and personal distress.
Patient Health | Baseline, 2-weeks
  A 2-item instrument using a 0-3 Likert (0 = not at all … 3 = nearly every day) that measures participants' perceived depression over the last 2-weeks.
Revised Self-Monitoring | Baseline, 2-weeks
  A 13-item instrument using a 1-5 Likert (1 = … 5 = ) to measure socioemotional sensitivity and responsiveness to the behavioral expressions of others. An example is "In conversations, the subject is sensitive to even the slightest change in the facial expression of the other person he/she is conversing with."
Self-Compassion | Baseline, 2-weeks
  A 12-item instrument using a 1-5 Likert (1 = almost never … 5 = almost always) to measure an individual's self-compassion. An example is "When I fail at something important to me I become consumed by feelings of inadequacy."
Inclusion of Self in Other | Baseline, 2-weeks
  A 7-item instrument using concentric circles (1 = no overlap … 7 = most overlap) to measure an individual's perceived relationship between self to other.

SECONDARY OUTCOMES:
Patient resting state functional connectivity (RSFC) | From date of completion of collection of all primary outcome measures, assessed up to 24 months
  Pre-gathered RSFC will be used in mixed models to determine its predictive potential on rhythm production, social attention, and connectedness.
Perceptions of relationship quality between participants as determined by word frequency analysis of semi-structured interview data | From date of completion of collection of all primary outcome measures, assessed up to 24 months
  Semi-structured interviews between participants of the dyad-pair will be analyzed using qualitative data analysis software for word frequencies of subjective and objective perceptions of their relationship with one another.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Colverson, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Sandler Neurosciences Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spinosa V, Vitulli A, Logroscino G, Brattico E. A Review on Music Interventions for Frontotemporal Aphasia and a Proposal for Alternative Treatments. Biomedicines. 2022 Dec 29;11(1):84. doi: 10.3390/biomedicines11010084. PMID 36672592
- [Background] Clarke E, DeNora T, Vuoskoski J. Music, empathy and cultural understanding. Phys Life Rev. 2015 Dec;15:61-88. doi: 10.1016/j.plrev.2015.09.001. Epub 2015 Sep 7. PMID 26419700
- [Background] Hobeika L, Ghilain M, Schiaratura L, Lesaffre M, Puisieux F, Huvent-Grelle D, Samson S. The effect of the severity of neurocognitive disorders on emotional and motor responses to music. Ann N Y Acad Sci. 2022 Dec;1518(1):231-238. doi: 10.1111/nyas.14923. Epub 2022 Nov 2. PMID 36321882
- [Background] Hobeika L, Ghilain M, Schiaratura L, Lesaffre M, Huvent-Grelle D, Puisieux F, Samson S. Socio-emotional and motor engagement during musical activities in older adults with major neurocognitive impairment. Sci Rep. 2021 Jul 27;11(1):15291. doi: 10.1038/s41598-021-94686-4. PMID 34315954
- [Background] Kumfor F, Honan C, McDonald S, Hazelton JL, Hodges JR, Piguet O. Assessing the "social brain" in dementia: Applying TASIT-S. Cortex. 2017 Aug;93:166-177. doi: 10.1016/j.cortex.2017.05.022. Epub 2017 Jun 7. PMID 28662418
- [Background] Colverson A, Barsoum S, Cohen R, Williamson J. Rhythmic musical activities may strengthen connectivity between brain networks associated with aging-related deficits in timing and executive functions. Exp Gerontol. 2024 Feb;186:112354. doi: 10.1016/j.exger.2023.112354. Epub 2024 Jan 3. PMID 38176601